CLINICAL TRIAL: NCT07407218
Title: The Effect Of Fecal Microbiota And Selected Metabolites On Efficacy And Toxicity Of Radiotherapy In Head And Neck Patients
Brief Title: Fecal Microbiota And Metabolites In Head And Neck Cancer Patients Receiving (Chemo)Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OI-LJ-HN-MICROBIOME-2021; ERIDSPRA-0087/2021 (Other: Ministry of Health of the Republic of Slovenia)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Cancer (H&N)
Keywords: Fecal Microbiome; Gut Microbiota
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-arm study. All participants receive standard radical (chemo)radiotherapy according to institutional clinical practice and international guidelines. Biological samples (stool and blood) are collected at predefined time points during treatment for microbiome and metabolomics analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radical (Chemo)Radiotherapy With Microbiome and Metabolite Assessment (Experimental): atients with locally advanced head and neck cancer treated with radical radiotherapy with or without concurrent chemotherapy will provide two stool samples and two additional blood samples (7 mL each) during the course of treatment. Stool samples will be analyzed for fecal microbiota composition using 16S rRNA gene sequencing (V3-V4 regions) and PCR quantification of butyrate-production genes (but and buk). Stool and serum samples will also be analyzed for short-chain fatty acids and tryptophan metabolites using liquid chromatography-mass spectrometry (LC-MS). Treatment response and acute toxicity will be assessed according to standard clinical practice.
  Interventions: Radiation: Radical (Chemo)Radiotherapy

INTERVENTIONS:
Radiation: Radical (Chemo)Radiotherapy — Participants receive standard radical radiotherapy for locally advanced head and neck cancer, with or without concurrent chemotherapy, according to institutional clinical practice and international guidelines. During treatment, additional stool and blood samples are collected for microbiome (16S rRNA sequencing, but/buk gene quantification) and metabolite analyses (short-chain fatty acids and tryptophan metabolites by LC-MS) to evaluate associations with treatment response and acute toxicity.

SUMMARY:
This clinical study investigates whether the composition of the fecal microbiome and selected bacterial metabolites are associated with the efficacy and acute toxicity of radiotherapy in patients with locally advanced head and neck cancer treated with radical (chemo)radiotherapy. Increasing evidence suggests that gut bacteria and their metabolites may influence treatment response and side effects of cancer therapies, including radiotherapy.

Participants will receive standard radical radiotherapy with or without concomitant chemotherapy according to clinical guidelines. During the course of treatment, participants will provide two stool samples and two blood samples. Stool samples will be collected at home and delivered to the hospital on the day of radiotherapy. Blood samples (7 ml) will be collected during routine clinical blood draws. Samples will be analyzed to determine fecal microbiome composition using 16S rRNA sequencing and quantification of butyrate-producing bacterial genes (buk and but), as well as concentrations of short-chain fatty acids and tryptophan metabolites using targeted metabolomics.

Clinical outcomes will include treatment response assessed by CT or PET-CT imaging 3 months after completion of therapy, acute toxicity (CTCAE v5.0), and follow-up survival outcomes. The study aims to identify microbiome-related biomarkers that may contribute to improved personalization of supportive interventions in the future.

DETAILED DESCRIPTION:
Head and neck cancer represents approximately 4-5% of all cancers worldwide and is associated with relatively poor survival outcomes. Most patients present with locoregionally advanced disease, and despite aggressive multimodal treatment including radiotherapy, recurrence occurs in up to half of patients within two years. Acute toxicities of radiotherapy, particularly radiomucositis and radiodermatitis, occur in more than 90% of patients and may lead to interruptions of treatment, negatively affecting outcomes.

Recent evidence indicates that the gut microbiome (fecal microbiota) and its metabolites may influence the efficacy and toxicity of cancer treatments. Studies have demonstrated associations between gut microbiota composition and response to immunotherapy and chemotherapy, and preclinical data suggest that specific bacterial metabolites, including short-chain fatty acids and tryptophan metabolites, may affect radiotherapy-related toxicity and survival. Emerging clinical studies have also shown associations between baseline gut microbiome diversity and survival or response to chemoradiotherapy in several cancer types. However, data regarding patients with head and neck cancer remain limited.

This prospective clinical study aims to evaluate the association between fecal microbiome composition and selected bacterial metabolites with treatment response and acute toxicity in patients with locoregionally advanced head and neck cancer undergoing radical radiotherapy with or without concomitant chemotherapy at the Institute of Oncology Ljubljana.

Participants will be treated according to standard institutional clinical practice and international guidelines. Biological samples will be collected at two time points during treatment: (1) from the start of radiotherapy until 7 days after initiation, but before administration of the first chemotherapy cycle (if applicable), and (2) during the last 7 days of radiotherapy. At each time point, participants will provide a stool sample (10-20 ml) collected at home and stored at 4°C until delivery to the hospital. Additionally, a 7 ml blood sample will be collected during routine clinical blood draws. Samples will be processed and stored at -80°C.

Microbiome analysis will be performed using sequencing of the V3-V4 regions of the 16S rRNA gene. Key bacterial genes involved in butyrate production (buk and but) will be quantified using PCR. Targeted metabolomics using liquid chromatography-mass spectrometry (LC-MS) will be performed to quantify short-chain fatty acids and tryptophan metabolites in stool and serum samples.

Clinical and demographic data will be collected for each participant, including dietary intake during the 24 hours prior to sampling, radiotherapy dose-volume parameters, acute and late toxicity assessed using CTCAE v5.0, and response to treatment assessed by CT or PET-CT imaging 3 months after completion of (chemo)radiotherapy according to RECIST 1.1 criteria. Participants will be followed for recurrence-free survival and overall survival for two years.

The primary outcome is treatment response, defined as complete response versus incomplete response at the 3-month imaging evaluation. Secondary outcomes include overall survival, recurrence-free survival at two years, and acute treatment-related toxicity. Statistical analyses will include assessment of alpha and beta diversity, PERMANOVA analysis, and logistic regression models to evaluate associations between microbiome characteristics, metabolite concentrations, and clinical outcomes.

The study is exploratory and designed as a signal-finding study. Based on comparable published studies and feasibility considerations, approximately 60 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years)

Carcinoma of the oral cavity, oropharynx, nasopharynx, hypopharynx, larynx, or carcinoma metastases in cervical lymph nodes of unknown primary origin

Overall stage III-IV according to the 8th TNM classification

Planned radical radiotherapy with or without concomitant chemotherapy

Exclusion Criteria:

Planned induction chemotherapy

Failure to complete radical (chemo)radiotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Treatment Response | 3 months after completion of (chemo)radiotherapy
  Response to treatment assessed within routine clinical practice by CT or PET-CT imaging 3 months after completion of (chemo)radiotherapy, comparing patients with complete response versus incomplete response
Treatment Response | 3 months after completion of (chemo)radiotherapy
  Response to treatment assessed within routine clinical practice by CT or PET-CT imaging 3 months after completion of (chemo)radiotherapy, comparing patients with complete response versus incomplete response.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No